CLINICAL TRIAL: NCT05266248
Title: Pilot Study Characterizing the Pharmacokinetic Profile of a Novel Encapsulated Caffeine Beverage in the Fed and Fasted States
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-2116
Record Dates: First submitted 2022-01-26; First posted 2022-03-04 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Pharmacokinetics
Keywords: caffeine; plasma; encapsulated; beverage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fed state (Experimental): Standardized high fat breakfast before dosing
  Interventions: Other: 250 mg encapsulated caffeine
- Fasted state (Experimental): Remain fasted for 4 hours post-dose
  Interventions: Other: 250 mg encapsulated caffeine

INTERVENTIONS:
Other: 250 mg encapsulated caffeine — Zero calorie 500 ml (16.9 oz) flavored, carbonated energy beverage

SUMMARY:
Pilot study designed to characterize the plasma caffeine pharmacokinetic profile of encapsulated caffeine when consumed in the fasted and fed states.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and female volunteers aged 18 to 55 years.
2. Have a BMI of 18 to 29.9 kg/m2 (inclusive)
3. Are regular caffeine consumers (average 1 to 3 caffeine-containing beverages per day, not to exceed 400 mg/ per day)
4. Willing to commit to 1 overnight stays (~36 hrs)
5. Able to comprehend and willing to sign an Informed Consent Form (ICF)
6. Willing to avoid caffeine-containing products for ≥48 hrs prior to dosing and until the completion of each test visit
7. Willing to avoid alcohol for ≥24 hrs prior to dosing
8. Willing to fast 10 hrs prior to dosing
9. Willing to stick to their usual dietary patterns and avoid grapefruit
10. Willing to stick to their usual physical activity level throughout the study
11. Willing to stick to their usual sleep pattern
12. Willing and able to consume a high-fat, high-caloric breakfast
13. No participation in any clinical trial within the past 30 days or 5 half lives and throughout this study, or any PEP protocol within the past 6 months.

Exclusion Criteria:

1. Reported history or clinical manifestations of significant metabolic (including type 1 or type 2 diabetes mellitus), hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, or psychiatric disorders unless deemed clinically not significant by investigator
2. Current or recent history (<30 days prior to Screening) of a clinically significant bacterial, fungal, or mycobacterial infection
3. Current clinically significant viral infection
4. History of malignancy within the past 5 years, with the exception of cured basal cell or squamous cell carcinoma of the skin within 6 months
5. Are pregnant or breastfeeding or planning to become pregnant
6. Resting heart rate less than 45 bpm or greater than 100 bpm.
7. History of unstable ischemic heart disease or uncontrolled hypertension (blood pressure 150/90 mm Hg)
8. History of significant surgery that may affect absorption of caffeine. Appendectomy and/or cholecystectomy will be allowed.
9. Presence of a malabsorption syndrome possibly affecting drug/Product absorption (e.g., Crohn's disease or chronic pancreatitis).
10. Extreme dietary habits, including but not limited to intentional consumption of a high fiber diet, gluten-free, low-carb, vegan, ketogenic.
11. History of alcoholism or drug addiction within 1 year prior to Screening, or current alcohol or drug use that, in the opinion of the investigator, will interfere with the subject's ability to comply with the dosing schedule and study evaluations.
12. More than one tobacco-containing or nicotine-containing product occasions per month on average, or use of such products within 48 hours prior to dosing of each study period
13. Use of any prescription or nonprescription drugs (including vitamins, minerals, and phytotherapeutic, herbal, or plant-derived preparations) is prohibited within 7 days prior to the dose of study product, unless deemed acceptable by the Investigator.
14. Use of any medication known to have an interaction with caffeine including oral contraceptives (e.g., medications metabolized via the CYP1A2 pathway). Contraceptives with localized effects (e.g., copper and hormonal IUDs, vaginal ring) are acceptable, methods with systemic effects (e.g., patch or subdermal implants/devices) are not.
15. Use of any medication known to alter the pH of the gastrointestinal tract (e.g., proton-pump inhibitors, histamine H2-receptor antagonists (H2 blockers), antacids, etc.).
16. Donation of blood in excess of 500 ml within 4 weeks prior to study entry or of plasma within 2 weeks prior to Screening.
17. Receipt of blood products within 3 months prior to study entry.
18. Subjects who, in the opinion of the investigator, are unable or unlikely to comply with the dosing schedule and study evaluations

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Area under the concentration curve for plasma caffeine (AUC0-t) | Changes from pre-dose to 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, and 6 hours after the first sip of beverage ingestion
  Plasma caffeine pharmacokinetics
Peak caffeine concentration (Cmax) | Changes from pre-dose to 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, and 6 hours after the first sip of beverage ingestion
  Plasma caffeine pharmacokinetics
Time to maximal plasma caffeine concentration (Tmax) | Changes from pre-dose to 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, and 6 hours after the first sip of beverage ingestion
  Plasma caffeine pharmacokinetics
Plasma caffeine concentration by time profile | Changes from pre-dose to 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, and 6 hours after the first sip of beverage ingestion
  Plasma caffeine pharmacokinetics

SECONDARY OUTCOMES:
Vital sign measurement: Systolic and diastolic blood pressure | Changes in systolic and diastolic blood pressure over 6.5 hours, from prior to blood sample collection at -30 minutes pre-dose to 2 and 6 hours after the first sip of beverage ingestion
  Safety parameter: Blood pressure
Vital sign measurement: Heart rate | Changes in heart rate over 6.5 hours, from prior to blood sample collection at -30 minutes pre-dose to 2 and 6 hours after the first sip of beverage ingestion
  Safety parameter: Heart rate
Occurrence of Adverse events | From the first sip of beverage ingestion (Time 0) of the first dosing day, until the subject exits the study the evening of the second and last dosing day. The two dosing days are approximately 7 days apart.
  Safety parameter: Treatment-emergent AEs (TEAEs) and adverse drug reactions (ADRs)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Galitz, MD, Principal Investigator — GCP, Global Clinical Professionals
Locations (1):
- GCP Research, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No